CLINICAL TRIAL: NCT02140021
Title: Prevalence of Anal Dysplasia and Anal Cancer in Women With Cervical, Vaginal and Vulvar Dysplasia and Cancer
Brief Title: Biospecimen Collection and Testing for the Prevalence of Anal Dysplasia and Anal Cancer in Patients With Cervical, Vaginal and Vulvar Dysplasia and Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2014-0021; NCI-2018-02553 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0021 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenocarcinoma In Situ; Cervical Intraepithelial Neoplasia; Cervical Squamous Cell Carcinoma, Not Otherwise Specified; Cervical Squamous Intraepithelial Neoplasia; Early Invasive Cervical Adenocarcinoma; Early Invasive Cervical Squamous Cell Carcinoma; High Grade Cervical Squamous Intraepithelial Neoplasia; High Grade Vaginal Intraepithelial Neoplasia; Low Grade Vaginal Intraepithelial Neoplasia; Stage I Cervical Cancer AJCC v8; Stage I Vaginal Cancer AJCC v8; Stage I Vulvar Cancer AJCC v8; Stage IA Cervical Cancer AJCC v8; Stage IA Vaginal Cancer AJCC v8; Stage IA Vulvar Cancer AJCC v8; Stage IA1 Cervical Cancer AJCC v8; Stage IA2 Cervical Cancer AJCC v8; Stage IB Cervical Cancer AJCC v8; Stage IB Vaginal Cancer AJCC v8; Stage IB Vulvar Cancer AJCC v8; Stage IB1 Cervical Cancer AJCC v8; Stage IB2 Cervical Cancer AJCC v8; Stage II Cervical Cancer AJCC v8; Stage II Vaginal Cancer AJCC v8; Stage II Vulvar Cancer AJCC v8; Stage IIA Cervical Cancer AJCC v8; Stage IIA Vaginal Cancer AJCC v8; Stage IIA1 Cervical Cancer AJCC v8; Stage IIA2 Cervical Cancer AJCC v8; Stage IIB Cervical Cancer AJCC v8; Stage IIB Vaginal Cancer AJCC v8; Stage III Cervical Cancer AJCC v8; Stage III Vaginal Cancer AJCC v8; Stage III Vulvar Cancer AJCC v8; Stage IIIA Cervical Cancer AJCC v8; Stage IIIA Vulvar Cancer AJCC v8; Stage IIIB Cervical Cancer AJCC v8; Stage IIIB Vulvar Cancer AJCC v8; Stage IIIC Vulvar Cancer AJCC v8; Stage IV Cervical Cancer AJCC v8; Stage IV Vaginal Cancer AJCC v8; Stage IV Vulvar Cancer AJCC v8; Stage IVA Cervical Cancer AJCC v8; Stage IVA Vaginal Cancer AJCC v8; Stage IVA Vulvar Cancer AJCC v8; Stage IVB Cervical Cancer AJCC v8; Stage IVB Vaginal Cancer AJCC v8; Stage IVB Vulvar Cancer AJCC v8; Vaginal Adenocarcinoma; Vulvar Adenocarcinoma; Vulvar High Grade Squamous Intraepithelial Lesion; Vulvar Intraepithelial Neoplasia; Vulvar Squamous Cell Carcinoma; Vulvar Squamous Intraepithelial Lesion
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening (biospecimen collection) (Experimental): Patients undergo collection of anal, cervical, vaginal, and oral samples during their scheduled pelvic exam.
  Interventions: Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo anal, cervical, vaginal, and oral sample collection
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This trial studies the prevalence of anal dysplasia and anal cancer in patients with cervical, vaginal, and vulvar dysplasia and cancer. Studying samples collected from patients in the laboratory may help doctors learn more about the human papillomavirus and how often anal cancer occurs in patients with cervix, vagina, or vulvar cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the prevalence of invasive squamous cell carcinoma of the anus in women with high-grade dysplasia or carcinoma of the cervix, vagina or vulva.

SECONDARY OBJECTIVES:

I. To estimate the prevalence of anal dysplasia in women with high-grade dysplasia or carcinoma of the cervix, vagina or vulva.

EXPLORATORY OBJECTIVES:

I. To estimate the clinical performance (sensitivity, specificity, positive and negative predictive values, and positive and negative likelihood ratios) of anal pap testing to diagnose anal dysplasia in women with high-grade dysplasia or carcinoma of the cervix, vagina or vulva.

II. To estimate the clinical performance (sensitivity, specificity, positive and negative predictive values, and positive and negative likelihood ratios) of anal high-risk human papillomavirus (HPV) testing to diagnose anal dysplasia in women with high-grade dysplasia or carcinoma of the cervix, vagina or vulva.

III. To estimate the clinical performance (sensitivity, specificity, positive and negative predictive values, and positive and negative likelihood ratios) of anal pap testing and HPV testing (anal "cotesting") to diagnose anal dysplasia in women with high-grade dysplasia or carcinoma of the cervix, vagina or vulva.

IV. To determine associations between gut and cervical microbiomes and anal dysplasia/carcinoma in women with high-grade dysplasia or carcinoma of the cervix, vagina, or vulva.

V. To estimate the prevalence of oral HPV infection in women with high-grade dysplasia or carcinoma of the cervix, vagina or vulva.

VI. To compare a new HPV point of care test developed by Rice University with current standard HPV testing.

OUTLINE:

Patients undergo collection of anal, cervical, vaginal, and oral samples during their scheduled pelvic exam.

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically confirmed cervical, vaginal or vulvar high-grade dysplasia, invasive squamous cell carcinoma, invasive adenocarcinoma, or adenocarcinoma-in-situ (AIS). All stages and grades will be eligible.
* Women with a diagnosis of high grade intraepithelial lesion (HSIL) from a routine pap test.
* Patients must sign an approved informed consent document.

Exclusion Criteria:

* Patients with previously documented perianal squamous cell dysplasia or invasive squamous cell carcinoma of the anus or anal canal.
* Patients unwilling or unable to provide informed consent for the study.
* Male patients will not be included in this study.
* Patients with previously documented HPV related oropharyngeal cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2014-10-27 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Prevalence of invasive squamous cell carcinoma of the anus | Up to 5 years
  Will estimate the prevalence of invasive squamous cell carcinoma of the anus in women with 95% confidence intervals.
Sensitivity and specificity of anal pap testing to diagnose anal dysplasia | Up to 5 years
  Will use the results of anoscopy as the true state of the patient and will estimate with 95% confidence intervals.
Sensitivity and specificity of anal human papillomavirus (HPV) testing to diagnose anal dysplasia | Up to 5 years
  Will use the results of anoscopy as the true state of the patient and will estimate with 95% confidence intervals.
Sensitivity and specificity of the combination of anal pap testing + anal HPV testing to diagnose anal dysplasia | Up to 5 years
  Will use the results of anoscopy as the true state of the patient and will estimate with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Schmeler, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas

DOCUMENTS (1):
  • Informed Consent Form (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/21/NCT02140021/ICF_000.pdf